CLINICAL TRIAL: NCT07262021
Title: Comparison of Visual Function of Enhanced Monofocal Intraocular Lenses After Cataract Surgery
Brief Title: Visual Function of Enhanced Monofocal Intraocular Lenses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Art25
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; intraocular surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art 25 IOL (Experimental): Patient will receive the Art 25 IOL during cataract surgery
  Interventions: Device: enhanced monofocal IOL
- Eyhance (Experimental): Patient will receive the Eyhance IOL during cataract surgery
  Interventions: Device: enhanced monofocal IOL

INTERVENTIONS:
Device: enhanced monofocal IOL — Art 25 IOL, enhanced monofocal IOL
  Arms: Art 25 IOL
Device: enhanced monofocal IOL — Eyhance IOL, enhanced monofocal IOL
  Arms: Eyhance

SUMMARY:
Comparison of the visual function of two enhanced monofocal intraocular lenses after cataract surgery

DETAILED DESCRIPTION:
Cataracts remain the leading cause of preventable blindness in many developing countries. Over the past decades, cataract surgery has undergone significant advancements. With the development of refined surgical techniques, such as smaller incisions, and the introduction of advanced intraocular lens (IOL) technologies, the procedure has transformed into a refractive approach for visual rehabilitation. The primary goal is to achieve a high level of spectacle independence for patient.

Monofocal lenses are designed with a single fixed focal length and refractive power. While they provide excellent distance vision, patients still need glasses for intermediate and near vision. However, modern patients have increasingly high expectations, often seeking full independence from spectacles after cataract surgery. This growing demand has fueled ongoing research and innovation in the development of advanced IOLs. In contrast, enhanced monofocal IOLs offer optical properties that deliver good intermediate vision outcomes without the negative aspects of multifocal IOLs such as photic phenomena or loss in contrast vision.

The aim of the study is therefore to compare two refractive enhanced monofocal IOLs in an intra-individual approach.

60 eyes of 30 patients will be included into this study. After randomization one eye is implanted with the Art 25 IOL, whereas the other eye gets the Eyhance IOL. Follow-up visits will be 1 week and 3 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* age-related bilateral cataract
* Age 21 or older
* Visual acuity > 0.05
* Axial length: 21.00-27.00mm
* Astigmatism < 1.0 dpt
* Normal findings in the medical history and physical examination
* Written informed consent prior to surgery

Exclusion Criteria:

* Reduced contrast vision, binocularity or stereoscopic vision (e.g. amblyopia, strabismus)
* Active ocular disease (e.g chronic uveitis, diabetic retinopathy, chronic glaucoma not responsive to medication, corneal dystrophies, etc.) precluding good post- operative visual acuity
* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome
* Irregular astigmatism on corneal tomography
* Pronounced dry eye disease
* Nystagmus or pathologies that might affect patient's fixation
* Previous ocular surgery or trauma
* Persons who are pregnant or nursing

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Distance-corrected intermediate visual acuity | 3 months
  The difference in distance-corrected intermediate visual acuity before and after surgery will be measured at 66 cm and compared between the two different IOLs

SECONDARY OUTCOMES:
Uncorrected intermediate visual acuity | 3 months
  The difference in uncorrected intermediate visual acuity before and after surgery will be measured at 66 cm and compared between the two different IOLs
Corrected and uncorrected distance visual acuity | 3 months
  The difference in corrected and uncorrected distance visual acuity before and after surgery will be measured at 4 m and compared between the two different IOLs
Corrected and uncorrected near visual acuity | 3 months
  The difference in corrected and uncorrected near visual acuity before and after surgery will be measured at 40 cm and compared between the two different IOLs
Defocus curve | 3 months
  The difference in visual acuity assessed in the defocus curve before and after surgery and compared between the two different IOLs
Contrast Sensitivity | 3 months
  The difference in contrast sensitivity between the two different IOLs

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Univ.-Prof. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided